CLINICAL TRIAL: NCT00267020
Title: A Randomized, Open-Label Phase 2 Study of 2 Regimens, Gemcitabine Plus Enzastaurin and Single-Agent Gemcitabine, in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Phase 2 Study of Gemcitabine or Gemcitabine + Enzastaurin in Participants With Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10463; H6Q-US-S002 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — enzastaurin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzastaurin+Gemcitabine (Experimental)
  Interventions: Drug: enzastaurin; Drug: gemcitabine
- Gemcitabine (Active Comparator)
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: enzastaurin — 1200 milligrams (mg) loading dose then 500 mg, orally, daily, six 28-day cycles
  Other Names: LY317615
  Arms: Enzastaurin+Gemcitabine
Drug: gemcitabine — 1000 milligrams/square meter (mg/m^2), intravenously on Days 1, 8 and 15 per cycle, six 28-day cycles
  Other Names: LY188011; Gemzar

SUMMARY:
The purpose of this research study is to determine the effects and toxicity of gemcitabine alone or gemcitabine plus enzastaurin in participants with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the pancreas.
* Pretreatment tumor specimen must be available.
* No prior chemotherapy immunotherapy, biological therapy, or hormonal therapy for pancreatic cancer, including 5-fluorouracil (5-FU) with radiation therapy.
* Prior radiation allowed.
* Ability to stop some types of anti-seizure medicines within 14 days of enrollment.

Exclusion Criteria:

* Endocrine pancreatic tumor or ampullary cancer.
* Central Nervous System (CNS) metastases.
* Inability to swallow tablets.
* 10% or greater weight loss over the 6 weeks before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Dallas, Texas, United States

REFERENCES:
- [Background] Yount S, Cella D, Webster K, Heffernan N, Chang C, Odom L, van Gool R. Assessment of patient-reported clinical outcome in pancreatic and other hepatobiliary cancers: the FACT Hepatobiliary Symptom Index. J Pain Symptom Manage. 2002 Jul;24(1):32-44. doi: 10.1016/s0885-3924(02)00422-0. PMID 12183093
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow reports those participants who discontinued from study drug.
Groups:
- Enzastaurin+Gemcitabine: Enzastaurin: 1200 milligrams (mg) administered orally (as three 400-mg doses) after a meal on Day 1, then 500 mg orally, daily (as five 100-mg tablets) after lunch on Days 2 to 28 in Cycle 1, then 500 mg orally, daily (as five 100-mg tablets) after lunch on Days 1 to 28 in Cycle 2 and later.
  Gemcitabine: 1000 milligrams/square meter (mg/m^2) administered intravenously on Days 1, 8 and 15 of each 28-day cycle.
- Gemcitabine: Gemcitabine: 1000 milligrams/square meter (mg/m^2) administered intravenously on Days 1, 8 and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine
Started | 86 | 44
Received at Least 1 Dose | 82 | 39
Per-Protocol Population | 81 (With: cancer of the pancreas;no other chemotherapy;disease at baseline;received 1 dose of study drug) | 38 (With: cancer of the pancreas;no other chemotherapy;disease at baseline;received 1 dose of study drug)
Completed | 0 | 1
Not Completed | 86 | 43
Not completed — Adverse Event | 22 | 5
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 17 | 7
Not completed — Physician Decision | 3 | 2
Not completed — Disease Progression | 39 | 25
Not completed — Unrelated Complication | 1 | 1
Not completed — Sponsor Request | 1 | 0
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All randomized participants.
Groups:
- Gemcitabine: Gemcitabine: 1000 mg/m^2 administered intravenously on Days 1, 8 and 15 of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine | Total
Number analyzed (Participants) | 86 | 44 | 130
Age, Continuous [Median (Full Range); unit: years] | 68.3 [39.6 to 86.7] | 64.1 [41.9 to 83.4] | 67.6 [39.6 to 86.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 12 | 52
  Male | 46 | 32 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12
  Not Hispanic or Latino | 77 | 41 | 118
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69 | 35 | 104
  Black or African American | 7 | 5 | 12
  Asian | 1 | 1 | 2
  Hispanic | 9 | 3 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86 | 44 | 130
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — [1] ECOG is a scale of participants activity Status 0 - Fully Active
  1. - Ambulatory, Restricted Strenuous Activity
  2. - Ambulatory, No Work Activities
  Participants
    0 - Fully Active | 36 | 16 | 52
    1 - Ambulatory, Restricted Strenuous Activity | 43 | 25 | 68
    2 - Ambulatory, No Work Activities | 7 | 3 | 10
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] | 1.8 (0.24) | 1.9 (0.21) | 1.8 (0.23)
Diagnosis Stage [Count of Participants; unit: Participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body).
  Stage IIA -The tumor is outside pancreas but not in large blood vessels or lymph nodes; Stage IIB: Cancer in or outside pancreas but not in large blood vessels; spread to nearby lymph nodes.
  Stage III - The tumor is outside pancreas and spread to nearby large blood vessels or major nerves. May or may not have spread to nearby lymph nodes; not spread to distant sites.
  Stage IV - the cancer has spread to other organs of the body such as the lung, brain, or liver.
  Participants
    Stage IIA | 3 | 0 | 3
    Stage IIB | 4 | 2 | 6
    Stage III | 7 | 7 | 14
    Stage IV | 72 | 35 | 107
Current Stage [Count of Participants; unit: Participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body).
  Stage IIB: Cancer in or outside pancreas but not in large blood vessels; spread to nearby lymph nodes.
  Stage III - The tumor is outside pancreas and spread to nearby large blood vessels or major nerves. May or may not have spread to nearby lymph nodes; not spread to distant sites.
  Stage IV - the cancer has spread to other organs of the body such as the lung, brain, or liver.
  Participants
    Stage IIB | 1 | 1 | 2
    Stage III | 7 | 5 | 12
    Stage IV | 78 | 38 | 116

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was the duration from randomization to death. OS was censored at the last contact for participants who were alive, at the cut-off date.
Time Frame: Randomization to the date of death from any cause up to 27.7 months
Population: Intent-to -treat (ITT) population: All randomized participants. Participants censored: Enzastaurin+Gemcitabine = 17; Gemcitabine = 11.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine
Number analyzed (Participants) | 86 | 44
months | 5.6 [4.2 to 6.9] | 5.1 [3.6 to 8.1]

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Response Rate)
Description: Response rate was defined as percentage of responders (best study response recorded as CR or PR) from the qualified number of participants for tumor response analysis. Response defined using Response Evaluation Criteria In Solid Tumors (RECIST, v1.0) criteria: CR was disappearance of all target lesions for at least 4 weeks. PR was at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of LD.
  Percentage of participants was calculated as: (The number of responders with CR or PR/ The number of participants qualified for tumor response analysis) × 100.
Time Frame: Randomization to measured progressive disease (PD) up to 19.9 months
Population: Per Protocol Population: Randomized participants who had: 1) histological or cytological diagnosis of locally advanced (Stage II, III) or metastatic (Stage IV) adenocarcinoma of the pancreas; 2) no concurrent systemic chemotherapy; 3) presence of measurable disease at baseline; and 4) received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine
Number analyzed (Participants) | 81 | 38
percentage of participants
  CR | 1.2 [0.0 to 6.7] | 0 [0 to 0]
  PR | 7.4 [2.8 to 15.4] | 5.3 [0.6 to 17.7]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the first date of documented progressive disease (PD) or death due to any cause, whichever occurred first. PFS was censored at the date of the last assessment visit for participants who were still alive at data cut-off and who had not had documented progressive disease. Participants who started a new treatment before progression were censored as of the date of the start of new treatment.
Time Frame: Randomization to measured PD or death from any cause up to 21.6 months
Population: Intent-to-treat (ITT) population: All randomized participants. Participants censored: Enzastaurin+Gemcitabine = 21; Gemcitabine = 10.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine
Number analyzed (Participants) | 86 | 44
months | 3.4 [2.4 to 4.0] | 3.0 [1.9 to 4.5]

4. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined, using the Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria, as the time from first objective status assessment of CR or PR to the first time of disease progression or death as a result of any cause. Using the Response Evaluation Criteria in Solid Tumors (RECIST V1.0) criteria, CR was defined as the disappearance of all tumor lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of LD. Duration of response was censored at the date of the last assessment visit for responders who were still alive at data cut-off and had no documented progressive disease (PD).
Time Frame: Time of response to PD or death from any cause up to 19.9 months
Population: Participants in the Per Protocol population with a CR or PR: With histological or cytological diagnosis of locally advanced adenocarcinoma of the pancreas; no concurrent systemic chemotherapy; presence of measurable disease at baseline; and treatment with at least 1 dose of study drug. Censored: Enzastaurin+Gemcitabine = 1; Gemcitabine = 0.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine
Number analyzed (Participants) | 7 | 2
months | 4.6 [3.7 to 13.9] | 9.2 [5.6 to 12.9]

5. Secondary Outcome: Change in Scores From Baseline (Improved, Stable or Worsened) to End of Study in Functional Assessment of Cancer Therapy Hepatobiliary Version 4 ( FACT-Hep v.4) (Quality of Life (QOL))
Description: FACT-Hep consists of 45 items in five subscales (1) physical well-being (PWB) score rage 0 -28; (2) social well-being (SWB) score range 0-28; (3) emotional well-being (EWB) score range 0-24; (4) functional well-being (FWB) score range 0-28; and (5) the hepatobiliary cancer subscale (HCS) Score range 0-72. The Trial Outcomes Index (TOI) is the sum of the PWB, FWB and Hep subscales with a scores range of 0 to 128. The Total FACT-Hep score was the sum of all questions with a scores range of 0 to 180. The Total FACT-G score was the sum of the 27 questions in the PWB, SFWB, EWB and FWB with a scores range of 0 to 108. The FACT-Hep Symptoms Index with 8 key questions and scores range of 0 to 32 from the Hep Subscale. Higher score in sub-score or total score indicates better QOL and better health state. Participants were classified as "Improved" if they had positive change from baseline, "Worsened" if they had negative change from baseline, and "Stable" otherwise.
Time Frame: Baseline through end of study up to 27.7 months
Population: All randomized participants who received at least one dose of study drug and had data for FACT-Hep questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine
Number analyzed (Participants) | 33 | 17
units on a scale
  Physical well-being- Improved: number analyzed (Participants) | 11 | 4
  Physical well-being- Improved | 7.2 (3.48) | 6.5 (2.71)
  Physical well-being- Stable: number analyzed (Participants) | 8 | 5
  Physical well-being- Stable | 0.3 (1.16) | 0.8 (1.80)
  Physical well-being- Worsened: number analyzed (Participants) | 14 | 8
  Physical well-being- Worsened | -10.0 (4.08) | -7.8 (3.96)
  Social well-being- Improved: number analyzed (Participants) | 7 | 5
  Social well-being- Improved | 3.8 (0.64) | 4.7 (2.10)
  Social well-being- Stable: number analyzed (Participants) | 20 | 8
  Social well-being- Stable | 0.1 (1.06) | -0.6 (1.21)
  Social well-being- Worsened: number analyzed (Participants) | 6 | 4
  Social well-being- Worsened | -6.5 (3.80) | -5.5 (2.66)
  Emotional well-being- Improved: number analyzed (Participants) | 8 | 3
  Emotional well-being- Improved | 6.9 (4.76) | 6.7 (3.79)
  Emotional well-being- Stable: number analyzed (Participants) | 14 | 9
  Emotional well-being- Stable | 0 (1.29) | -0.1 (1.36)
  Emotional well-being- Worsened: number analyzed (Participants) | 10 | 5
  Emotional well-being- Worsened | -5.8 (2.57) | -8.2 (4.15)
  Functional well-being- Improved: number analyzed (Participants) | 5 | 4
  Functional well-being- Improved | 6.8 (3.63) | 6.5 (1.73)
  Functional well-being- Stable: number analyzed (Participants) | 12 | 7
  Functional well-being- Stable | -0.2 (1.40) | -1.1 (0.90)
  Functional well-being- Worsened: number analyzed (Participants) | 15 | 6
  Functional well-being- Worsened | -10.6 (5.37) | -8.5 (4.42)
  Hepatobiliary cancer subscale- Improved: number analyzed (Participants) | 8 | 4
  Hepatobiliary cancer subscale- Improved | 12.7 (4.67) | 12.0 (5.20)
  Hepatobiliary cancer subscale- Stable: number analyzed (Participants) | 12 | 9
  Hepatobiliary cancer subscale- Stable | 0.5 (3.00) | 0.7 (3.78)
  Hepatobiliary cancer subscale- Worsened: number analyzed (Participants) | 12 | 4
  Hepatobiliary cancer subscale- Worsened | -14.6 (4.70) | -10.0 (4.32)
  Total Outcome Index- Improved: number analyzed (Participants) | 8 | 5
  Total Outcome Index- Improved | 21.4 (11.20) | 19.0 (11.49)
  Total outcome index- Stable: number analyzed (Participants) | 13 | 6
  Total outcome index- Stable | -1.6 (5.40) | -1.3 (4.76)
  Total outcome index- Worsened: number analyzed (Participants) | 11 | 6
  Total outcome index- Worsened | -35.9 (13.03) | -23.0 (9.88)
  Total FACT-Hep score- Improved: number analyzed (Participants) | 7 | 4
  Total FACT-Hep score- Improved | 30.0 (16.81) | 27.5 (17.91)
  Total FACT-Hep score- Stable: number analyzed (Participants) | 13 | 6
  Total FACT-Hep score- Stable | -1.2 (5.65) | 0 (4.19)
  Total FACT-Hep score- Worsened: number analyzed (Participants) | 12 | 7
  Total FACT-Hep score- Worsened | -37.9 (13.71) | -26.6 (12.26)
  Total FACT-G-score- Improved: number analyzed (Participants) | 7 | 2
  Total FACT-G-score- Improved | 19.1 (11.63) | 24.1 (18.95)
  Total FACT-G-score- Stable: number analyzed (Participants) | 9 | 7
  Total FACT-G-score- Stable | -0.5 (3.56) | -0.6 (4.17)
  Total FACT-G-score- Worsened: number analyzed (Participants) | 16 | 7
  Total FACT-G-score- Worsened | -20.1 (10.59) | -21.2 (10.75)
  FACT Hep Symptoms Index- Improved: number analyzed (Participants) | 13 | 6
  FACT Hep Symptoms Index- Improved | 7.4 (3.95) | 6.3 (2.50)
  FACT Hep Symptoms Index- Stable: number analyzed (Participants) | 5 | 7
  FACT Hep Symptoms Index- Stable | 0.5 (1.45) | 0.1 (1.85)
  FACT Hep Symptoms Index- Worsened: number analyzed (Participants) | 14 | 4
  FACT Hep Symptoms Index- Worsened | -7.0 (3.31) | -7.0 (2.16)

6. Secondary Outcome: Relationship of Steady-State Drug Levels to Clinical Outcomes of Overall Survival (OS)
Description: OS was the duration from randomization to death from any cause. For participants who were alive at data cut-off, OS was censored at the last contact. Participants were categorized into 2 groups based on their steady state drug levels of Enzastaurin (total analyte=enzastaurin + LSN326020 [metabolite]): those participants below the median and those participants above the median [2786.042 nanomoles per /liter (nmol/l)]. The steady state drug levels and clinical outcomes were not evaluated for the Gemcitabine only treatment group.
Time Frame: Randomization to date of death from any cause up to 27.7 months
Population: All participants who received at least 1 dose of study drug. Participants censored: Below median = 4; Above median =4.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin+Gemcitabine
Number analyzed (Participants) | 57
months
  Below median: number analyzed (Participants) | 29
  Below median | 7.2 [5.1 to 10.6]
  Above median: number analyzed (Participants) | 28
  Above median | 5.6 [3.2 to 6.9]

7. Secondary Outcome: Relationship of Steady-state Drug Levels to Best Overall Response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) (Disease Control)
Description: The overall disease control rate was calculated as percent of participants with overall response of complete response (CR), partial response (PR) or stable disease (SD) over number of per-protocol population. Using the Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria, CR: disappearance of all target and non-target lesions; PR: as at least a 30% decrease in sum of longest diameter (LD) of target lesions; progressive disease (PD) was defined as at least 20% increase in sum of LD of target lesions; SD: small changes that did not meet above criteria.
  Participants were categorized into 2 groups based on their steady state drug levels of Enzastaurin (total analyte=enzastaurin + LSN326020 [metabolite]): participants below the median and participants above the median [2754.521 nanomoles per liter (nmol/l)].
  The steady state drug levels and clinical outcomes were not evaluated for the Gemcitabine only group.
Time Frame: Beginning of treatment up to 27.7 months
Population: Randomized participants who had: 1) Histological or cytological diagnosis of locally advanced (Stage II, III) or metastatic (Stage IV) adenocarcinoma of the pancreas; 2) no concurrent systemic chemotherapy; 3) presence of measurable disease at baseline; and 4) received at least 1 dose of study drug and had data for overall response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin+Gemcitabine
Number analyzed (Participants) | 28
percentage of participants
  CR (Below median) | 3.6 [0.1 to 18.3]
  CR (Above median) | 0.0 [0.0 to 0.0]
  PR (Below median) | 17.9 [6.1 to 36.9]
  PR (Above median) | 3.6 [0.1 to 18.3]
  SD (Below median) | 57.1 [37.2 to 75.5]
  SD (Above median) | 39.3 [21.5 to 59.4]
  PD (Below median) | 14.3 [4.0 to 32.7]
  PD (Above median) | 32.1 [15.9 to 52.4]
  Disease Control (Below median) | 78.6 [59.0 to 91.7]
  Disease Control (Above median) | 42.9 [24.5 to 62.8]

8. Secondary Outcome: Carbohydrate Antigen 19-9 (CA 19-9) Concentration in the Blood
Description: CA19-9 is a tumor biomarker which was measured in the blood to assess the effect of treatment with enzastaurin.
Time Frame: Cycles 1 to 6, and post-treatment (up to 27.7 months)
Population: Safety population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: kilo units/liter (kU/L)
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine
Number analyzed (Participants) | 82 | 39
kilo units/liter (kU/L)
  Cycle 1 | 31708.5 (134178.00) | 12038.6 (26659.50)
  Cycle 2 | 12828.4 (33051.54) | 40764.9 (143995.67)
  Cycle 3 | 24709.5 (114098.20) | 1573.0 (2811.74)
  Cycle 4 | 37261.0 (168939.81) | 1102.7 (1547.67)
  Cycle 5 | 392.3 (744.91) | 403.1 (541.91)
  Cycle 6 | 600.9 (1268.90) | 938.5 (1542.34)
  Post-treatment 1st visit | 19420.5 (45867.95) | 11351.3 (23890.66)
  Post-treatment 2nd visit | 19557.7 (32615.58) | 93955.9 (176684.42)

9. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs) and Adverse Events (AEs) (Toxicity)
Description: Clinically significant events were defined as SAEs and other non-serious adverse events (AEs). Participants who died due to progressive disease (PD), AEs while on treatment or died during the 30 day post-treatment are included. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through study completion (Up To 27.7 Months)
Population: Safety population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine
Number analyzed (Participants) | 82 | 39
Participants
  Non-serious AEs | 80 | 38
  SAEs | 49 | 23
  Deaths due to PD | 3 | 1
  Deaths due to AEs | 4 | 1
  Deaths within 30-days after treatment | 3 | 1

ADVERSE EVENTS:
Time Frame: Baseline through study completion (27.7 months)
Description: Study-specific clinical outcomes due to progressive disease were not considered to be serious adverse events (SAEs) unless it was deemed related to study drug by the investigator.
Groups:
- Gemcitabine: Gemcitabine: 1000 mg/m^2 administered intravenously on Days 1, 8 and 15 of each of each 28-day cycle.
Arm/Group | Enzastaurin+Gemcitabine | Gemcitabine
Serious Adverse Events (participants affected / at risk) | 49/82 | 23/39
Other Adverse Events (participants affected / at risk) | 80/82 | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin+Gemcitabine (N=82) | Gemcitabine (N=39)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 3 (3)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Internal fixation of fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 5 (5)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin+Gemcitabine (N=82) | Gemcitabine (N=39)
Leukopenia (Blood and lymphatic system disorders) | 26 (26) | 14 (14)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Vision blurred (Eye disorders) | 2 (2) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 26 (26) | 8 (9)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 24 (24) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 25 (25) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 35 (35) | 13 (13)
Oesophagitis (Gastrointestinal disorders) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 17 (17) | 7 (7)
Chills (General disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 50 (50) | 22 (22)
Oedema (General disorders) | 10 (10) | 1 (1)
Oedema peripheral (General disorders) | 25 (25) | 12 (12)
Pain (General disorders) | 5 (5) | 3 (3)
Pyrexia (General disorders) | 15 (15) | 6 (6)
Hyperbilirubinaemia (Hepatobiliary disorders) | 7 (7) | 3 (3)
Hypersensitivity (Immune system disorders) | 2 (2) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Skin infection (Infections and infestations) | 4 (4) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 10 (10) | 6 (6)
Blood creatinine increased (Investigations) | 5 (5) | 1 (1)
Haemoglobin decreased (Investigations) | 46 (46) | 23 (23)
Laboratory test abnormal (Investigations) | 5 (5) | 1 (1)
Neutrophil count decreased (Investigations) | 32 (32) | 18 (18)
Platelet count decreased (Investigations) | 46 (46) | 20 (20)
Weight decreased (Investigations) | 9 (9) | 6 (6)
Weight increased (Investigations) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 23 (23) | 16 (16)
Dehydration (Metabolism and nutrition disorders) | 9 (9) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (9) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 (10) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4)
Ataxia (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 10 (10) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 6 (6) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6) | 3 (3)
Speech disorder (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (6) | 3 (3)
Depressed mood (Psychiatric disorders) | 8 (8) | 2 (2)
Insomnia (Psychiatric disorders) | 12 (12) | 2 (2)
Chromaturia (Renal and urinary disorders) | 10 (10) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Haematoma (Vascular disorders) | 6 (6) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 7 (7) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days